CLINICAL TRIAL: NCT06433739
Title: Efficacy of a Clinical Algorithm for the Selection of Peripheral Venous Catheters to Reduce the Number of Catheter-Associated Complications in Hospitalized Patients: A Retrospective Cohort Study
Brief Title: Efficacy of a Clinical Algorithm for the Selection of Peripheral Venous Catheters
Acronym: EACEC
Status: Completed | Type: Observational
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Other Study IDs: CSAPG-47
Record Dates: First submitted 2024-05-21; First posted 2024-05-30 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Catheter Related Complication
Keywords: Catheterization, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- appropriate catheter type selection: This group will include all peripheral venous catheterizations for which the appropriate catheter type selection according to the standardized algorithm has been performed
  Interventions: Other: standardized algorithm
- inappropriate catheter type selection: This group will include all peripheral venous catheterizations for which an inappropriate catheter type selection according to the standardized algorithm has been performed
  Interventions: Other: standardized algorithm

INTERVENTIONS:
Other: standardized algorithm — standardized algorithm for the correct selection of peripheral venous catheters

SUMMARY:
The aim of this observational study is to investigate the complications associated with peripheral venous catheterization based on whether a correct or incorrect catheter was used according to a clinical algorithm in patients admitted to an acute care unit. The main question it seeks to answer is:

• Are there fewer complications associated with catheterization when a correct catheter choice is made? Data from patients admitted to the acute care units of the sponsoring study center will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to acute care hospital wards.
* Carriers of a peripheral venous catheter.
* With the study evaluation criteria documented in their medical records.

Exclusion Criteria:

* Admitted to gynecology, obstetrics, and pediatrics wards.
* Admitted to the emergency department and intensive care units

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to some acute care unit requiring peripheral venous catheterization
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Catheters removed due to complications associated with the use of a peripheral venous catheter | Through study completion, an average of 1 year
  Percentage of catheters removed due to complications associated with the use of a peripheral venous catheter

SECONDARY OUTCOMES:
Selection of the peripheral venous catheter | Through study completion, an average of 1 year
  Correct or incorrect selection of the catheter according to the clinical algorithm. The proportion of correctly selected catheters in relation to the total number of catheters will be calculated.
Complications associated with the use of a peripheral venous catheter | Through study completion, an average of 1 year
  Number of complications associated with the use of a peripheral venous catheter depending on whether a correct or incorrect selection of the catheter was made according to the clinical algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Moreno, Principal Investigator — CSAPG
Locations (1):
- Consorci Sanitari Alt Penedes i Garraf, Sant Pere de Ribes, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.